CLINICAL TRIAL: NCT01745783
Title: Clinical Trial Phase I / II Multicenter, Randomized, Crossover, Double-blind Evaluation of the Safety and Feasibility of Systemic Therapy With Mesenchymal Cells Derived From Autologous Bone Marrow in Patients With Multiple Sclerosis
Brief Title: Mesenchymal Cells From Autologous Bone Marrow, Administered Intravenously in Patients Diagnosed With Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CeTMMo/EM/2010; 2010-023368-42 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-10 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Receive a single IV administration of cellular product (Bone marrow mesenchymal stem cells autologous) on Day 0 and placebo infusion on day + 180.
  Dose: 1-2x10^6 cells/Kg
  Interventions: Other: Bone marrow mesenchymal stem cells autologous
- Placebo Comparator (Placebo Comparator): Receive a placebo infusion on day 0 and a single administration cellular product on day +180. Dose: 1-2x10^6 cells/Kg
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Other: Bone marrow mesenchymal stem cells autologous — Infusion of mesenchymal cells from autologous bone marrow in a dose of 1-2x106 cells / kg
  Arms: Experimental
Other: Placebo comparator — Lactated Ringer's solution, 2.5% glucose and 1% human albumin.
  Arms: Placebo Comparator

SUMMARY:
This is a phase I / II for the evaluation of the safety and feasibility of intravenous infusion of mesenchymal cells from autologous bone marrow in patients with Multiple Sclerosis.

Intravenous administration of autologous mesenchymal cells of bone marrow is feasible and safe and can be effective in treating patients suffering from multiple sclerosis.

DETAILED DESCRIPTION:
The study population will consist of a total of 30 patients diagnosed with multiple sclerosis, who meet all inclusion criteria and none of the exclusion set and express their agreement to participate in the study by signing the informed consent of those whose results can be clinically evaluable.

Selected patients who consent will be enrolled in the trial and randomized to one of the following groups:

* Group 1 receiving a single intravenous administration of cellular product on Day 0 and placebo infusion on day + 180.
* Group 2 receiving a placebo infusion on day 0 and a single cell product administration on day +180.

Randomization will be 1:1, so that 15 patients will receive the cellular product on Day 0 (Group 1) and 15 patients on day +180 (group 2), always maintaining at all times the double-blind status of the test (patients and researchers).

The bone marrow will be extract from all patients immediately after inclusion in the study, under local anesthesia with sedation. For patients in group 1 autologous mesenchymal cells will be obtained from the bone marrow and infuse immediately after the time necessary for their production. For patients in group 2, bone marrow cells will be frozen for later procedure of mesenchymal cells and their infusion after six months.

Patients will be evaluated by clinical, radiological, and electrophysiological as well as detailed in section 8 corresponding to Development Test and Evaluation of Response.

It is estimated that the inclusion period is approximately 12-18 months, and each patient tracking another twelve months. Therefore the total duration of the study will be about 24 to 30 months from the inclusion of the first patient to completion follow-up period of the last patient included.

Study objectives:

* Main objectives: 1. To evaluate the safety of intravenous infusion of autologous bone marrow mesenchymal cells in multiple sclerosis patients diagnosed by evaluating complications and adverse effects of the therapy itself and study procedures.

  2. Assessing the difference in the number of lesions on magnetic resonance image with gadolinium, between the groups undergoing treatment at weeks 4, 12 and 24.
* Secondary objectives: 1. To evaluate the feasibility and efficacy of the indication of the treatment by analysis comparative results and exploratory clinical variables of patients at baseline (pretreatment) and at 6 and 12 months follow-up.

  2. Compare the results of safety, feasibility and efficacy between the administration initial cell therapy treatment (day 0) and that delayed (day +180).

  3. Evaluating the immunomodulatory effect of treatment by quantifying cell subsets and cytokines, functional analysis of the immune response. Cerebrospinal fluid metabolomic profile of gene expression of the cells present in blood and cerebrospinal fluid, with the aim of identifying new biomarkers with diagnosis of interest, prognosis or monitoring, and potential therapeutic targets that can be derived from it.

  4. Providing our results to the study proposed by the International Mesenchymal Stem Cell Transplant Study Group under whose directives will be performed the test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MS in their inflammatory forms :

1. Course outbreaks ( relapsing- remitting ) , who have not responded to at least one year of treatment with one or more of the approved therapies (beta - interferon, glatiramer acetate, natalizumab , mitoxantrone, fingolimod ) , confirmed by one or more of the following criteria:

   ( ii ) At least one clinically documented outbreak in the past 12 months. ( iii ) At least two clinically documented outbreaks in the last 24 months ( iv ) At least one lesion with gadolinium on MRI performed in the last 12 months.

   b . Secondary progressive forms that have not responded to at least one year of treatment with one or more of the approved therapies ( interferon beta , glatiramer acetate, natalizumab , mitoxantrone, fingolimod ) . That meet the following criteria:

   ( i ) Increase of 1 point or more if baseline EDSS score is less than or equal to 5.0 , or 0.5 point increase if the baseline score is greater than or equal to 5.5, in the last 12 months.

   ( ii ) at least one clinically documented outbreak or at least one lesion with gadolinium on MRI within the last 12 months.

   c . Primary progressive forms that meet the following three criteria:

   ( i ) Increase of 1 point or more if baseline EDSS score is less than or equal to 5.0 , or 0.5 point increase if the baseline score is greater than or equal to 5.5, in the last 12 months.

   ( ii ) At least 1 lesion with gadolinium on MRI within the last 12 months. ( iii ) oligoclonal bands in cerebrospinal fluid (CSF) .

   2 . Normal laboratory parameters , defined by:
   * Leukocytes ≥ 3000
   * Neutrophils ≥ 1500
   * Platelets ≥ 100,000
   * Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) ≤ 2.5 standard range institution
   * Creatinine ≤ 2.5 mg / dl

     3 . Patients of both sexes aged between 18 and 50.

     4 . Disease duration ≥ 2 years and ≤ 10 years.

     5 . EDSS (Expanded Disability Status Scale) between 3.0 and 6.5 points.

     6. Patients give their informed consent for participation in the clinical trial consent.

     7. Women of childbearing potential must have negative results on a pregnancy test at the time of inclusion in the study and agree to use a medically approved method of contraception while on study

   Exclusion Criteria:
   1. Any active or chronic infection, including Hepatitis B virus (HBV), Hepatitis C virus (HCV) or HIV .
   2. Immunosuppressive therapy in the 3 months prior to randomization (including natalizumab and fingolimod ).
   3. Treatment with interferon beta or glatiramer acetate in the 30 days prior to randomization .
   4. Corticosteroid therapy in the 30 days prior to randomization.
   5. Time since last exceeding 60 days prior to randomization outbreak.
   6. History of malignancy ( basal cell carcinoma of skin and carcinoma in situ are excluded in remission for over a year).
   7. Life expectancy severely limited by other co - morbidities.
   8. Previous history of myelodysplasia or hematological disease , or clinically relevant changes currently in the leukocyte count.
   9. Pregnancy / risk of pregnancy (including refusal to use contraception)
   10. Renal failure (eGFR <60 mL/min/1.37m2)
   11. Inability to undergo MRI scans
   12. Inability to give written informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Absence of unexpected serious adverse reactions as a measure of safety and reduction in number and volumes of the lesions on magnetic resonance image | 12 months

SECONDARY OUTCOMES:
Differences the results obtained in the two groups of patients due to determined parameters. | 12 months
  Secondary variables consist of differences the results obtained in the two groups of patients (treated versus treated at day 0 to day +180) at 12 month follow-up with respect to the following parameters:
  1. Disease activity on magnetic resonance (used one single combined index activity consisting of the presence of new or enlarged T2 or new or recurrence of injury).
  2. Changes in Expanded Disability Status Scale (EDSS).
  3. Changes Multiple Sclerosis Functional Composite (MSFC).
  4. Changes in quality of life scales
  5. Outbreaks: number and proportion of time off outbreaks.
  6. Disease-free patients (no sprouts, no progression and no activity in the RM).

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Izquierdo, MD, Principal Investigator — Section Chief of Neurology, University Hospital Virgen Macarena, Spain; Eduardo Agüera, MD, Principal Investigator — Section of Neurology, University Hospital Reina Sofía, Spain; Victoria Fernández, MD, Principal Investigator — Section of Neurophysiology, University Regional Hospital Carlos Haya, Spain; Inmaculada Concepción Herrera, MD, Study Chair — Technical Director of the Cell Therapy Unit, University Hospital Reina Sofia, Spain
Locations (3):
- Spain (3):
  - University Hospital Reina Sofia, Córdoba
  - University Regional Hospital Carlos Haya, Málaga
  - University Hospital Virgen Macarena, Seville

REFERENCES:
- [Derived] Uccelli A, Laroni A, Brundin L, Clanet M, Fernandez O, Nabavi SM, Muraro PA, Oliveri RS, Radue EW, Sellner J, Soelberg Sorensen P, Sormani MP, Wuerfel JT, Battaglia MA, Freedman MS; MESEMS study group. MEsenchymal StEm cells for Multiple Sclerosis (MESEMS): a randomized, double blind, cross-over phase I/II clinical trial with autologous mesenchymal stem cells for the therapy of multiple sclerosis. Trials. 2019 May 9;20(1):263. doi: 10.1186/s13063-019-3346-z. PMID 31072380
- See also: Andalusian Molecular Biology and Regenerative Medicine Centre — http://www.cabimer.es